CLINICAL TRIAL: NCT01912638
Title: Comparative Study of the Efficacy and Safety of Ologen Collagen Implant Versus Cohesive Viscoelastic in Trabeculectomy Performed for Steroid Induced Glaucoma
Brief Title: Trabeculectomy With Ologen Collagen Implant vs Trabeculectomy With Provisc in Steroid Induced Glaucoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Centre of Ophthalmology named after academician Zarifa Aliyeva (Other Government)
Collaborators: Aeon Astron Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trab-Olo-SG
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2015-07

CONDITIONS: Steroid Induced Glaucoma
Keywords: Trabeculectomy; Glaucoma; Steroids; Ologen; Viscoelastic
MeSH Terms: conditions — Glaucoma | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Implantation of Ologen in trabeculectomy (Experimental): Ologen Collagen Matrix is implanted in primary limbal-based trabeculectomy. It should be placed on the top of the loosely-sutured scleral flap before suturing of the conjunctiva thus preventing the collapse of the subconjunctival space.
  Interventions: Device: Ologen Collagen Matrix
- Provisc in trabeculectomy (Active Comparator): Provisc is used in primary limbal-based trabeculectomy. At the end of the surgery cohesive viscoelastic (Provisc) is injected under the scleral flap to prevent early hypotony.
  Interventions: Drug: Provisc

INTERVENTIONS:
Device: Ologen Collagen Matrix — Ologen is a porous collagen-glycosaminoglycan matrix that decrease early postoperative scarring after penetrating anti-glaucomatous surgery by randomized collagen deposition and microcyst formation. Implantation of Ologen Collagen Matrix in trabeculectomy was performed.
  Arms: Implantation of Ologen in trabeculectomy
Drug: Provisc — Provisc is an cohesive viscoelastic.
  Arms: Provisc in trabeculectomy

SUMMARY:
The purpose of this prospective randomized study is to assess and compare the clinical efficacy and safety of primary trabeculectomy with Ologen® collagen implant and cohesive viscoelastic (Provisc®) - augmented trabeculectomy in patients with medically uncontrolled steroid induced glaucoma.

DETAILED DESCRIPTION:
Steroid induced glaucoma is a well known and widely described disastrous clinical condition. However the subject of selection of most effective and safe treatment modality is still being discussed.

Sihota R et al reported that 26.5% cases required surgical treatment to control IOP. Unfortunately survival rate of successful blebs in 10 years after trabeculectomy varies from 40% to 60%. Anti-fibrotic agent MMC as adjunct to filtration surgery was used to prevent postoperative scarring that could compromise surgical success of trabeculectomy. Additional use of MMC in trabeculectomy leads to low final IOP but could be associated with such complications as cataract formation, intraocular toxicity, avascular filtering blebs, wound leakage, subsequent blebitis and endophthalmitis. Tissue-engineered biodegradable and biocompatible implant Ologen® Collagen Matrix may be used as an alternative to MMC. Ologen® is CE Mark and FDA approved artificial porcine extracellular matrix for modulating wound healing. Ologen® has been tested in animal models and has triple action:

1. prevent the collapse of the subconjunctival space;
2. guides the fibroblast to grow through the matrix pores thus preventing scar formation;
3. may act as an aqueous reservoir (avoids post-op hyperfiltration and shallow anterior chamber).

The filtering blebs scoring was performed by using Moorfields Bleb Grading System and Visante anterior segment optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years (inclusive)
* Patients with medically uncontrolled steroid induced glaucoma

Exclusion Criteria:

* Primary open angle glaucoma, angle-closure glaucoma, post-traumatic, uveitic, neovascular, or dysgenetic glaucoma
* Known allergic reaction to porcine collagen
* Preliminary conjunctival damage (trauma, vitreo-retinal surgery, previous glaucoma or strabismus surgery, etc)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | 2 years
  The absolute success was defined as an IOP less than 21 mmHg with no glaucoma medications.
  Follow-up visits were and will arranged at 1 and 2 first weeks, then every month during first 6 months, then every 3 months during 2.5 years after surgery.

SECONDARY OUTCOMES:
Postoperative complications | 2 years
  Complications were defined as follows: hypotony,shallow anterior chamber,serous or hemorrhagic choroidal detachment, hyphema,anterior chamber inflammation,persistent hypotonus maculopathy,corneal epithelial toxicity, "snuff" syndrome,blebitis or endophthalmitis,formation of Tenon's cyst.
Corrected distance visual acuity (CDVA) | 2 years
Appearance of the filtering bleb (FB) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elmar Kasimov, Professor, Study Director — Director of National Centre of Ophthalmology; Fidan Aghayeva, MD, Principal Investigator — Glaucoma consultant at National Centre of Ophthalmology
Locations (1):
- National Centre of Ophthalmology named after academician Zarifa Aliyeva, Baku, Azerbaijan

REFERENCES:
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740